CLINICAL TRIAL: NCT01978392
Title: MANAGE AT WORK: Evaluation of a Group-based Self-management Program to Address Workplace Discomfort and Fatigue Associated With Chronic Physical Health Conditions
Brief Title: MANAGE AT WORK: Addressing the Challenge of Chronic Physical Health Conditions in the Workplace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liberty Mutual Research Institute for Safety (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LMRIS 11-08; LMRIS Project 11-08 (Other Grant/Funding Number: Liberty Mutual Research Institute for Safety)
Record Dates: First submitted 2013-11-01; First posted 2013-11-07 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Chronic Physical Health Conditions
Keywords: disability; self-management; chronic illness; chronic pain; occupation; > 6 months
MeSH Terms: conditions — Chronic Disease; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-management group workshops (Experimental): Self-management group workshops: Participants randomized to the intervention arm will be asked to participate in group workshop sessions (10 hours total) led by a specially trained facilitator and provided over a span of approximately 2-3 months.
  Interventions: Behavioral: Self-management group workshops
- No treament (wait-list control) (No Intervention): Wait-list control: Participants randomized to the control arm will receive no intervention during the one-year period of data collection, but they will be invited to attend a full-day Saturday workshop after all study data collection is complete). The intent of the full-day workshop will be to provide the same self-management information as in the intervention arm, but on a delayed basis and in a more condensed format.

INTERVENTIONS:
Behavioral: Self-management group workshops — This intervention consists of multiple group workshop sessions (10 hours total) led by a specially trained facilitator and provided over a span of approximately 2-3 months. The intervention incorporates standard elements of existing evidence-based pain and illness self-management efforts, but tailoring key messages and discussion elements to apply to workplace problems most relevant to workers with chronic medical conditions. Each session is focused on different self-management strategies, with each session containing a mix of facilitator presentation, group discussion, case illustrations, role-play, completion of in-session self-assessments and activities, and brief homework assignments. Approximately equal time is allocated to the topics of improving comfort, modifying work, communicating effectively, applying systematic problem-solving strategies, and dealing with negative thoughts and emotions.
  Arms: Self-management group workshops

SUMMARY:
The specific aim of the study is to evaluate the health benefits of a series of group workshops designed for workers with chronic physical health conditions. The facilitated workshops apply principles of pain and illness self-management to help workers deal with health-related challenges while at work. The workshops address issues of pain management, physical job demands, pacing of work, communication, problem solving, and coping. Half of the participants in the study will be randomly assigned to attend workshop sessions (10 hours total), and all study participants will be followed for one year. The primary hypothesis is that workers who participate in these workshops will show improvements in work engagement and reductions in work limitation in the subsequent 12 months.

DETAILED DESCRIPTION:
One significant trend in the US workforce is the advancing median age of workers and the growing prevalence of chronic medical conditions that contribute to workplace pain, fatigue, task limitations, and reduced productivity. The proposed multi-site study is a randomized, controlled trial of a multi-session group intervention program targeting workers with chronic health concerns (N = 300). The primary outcome measures will be self-report measures of work limitations and work engagement measured at baseline, 6 months, and 12 months follow-up. Secondary outcomes will include turnover intention, sickness absence, job satisfaction, and healthcare utilization. Process variables and covariates will include assessment of self-efficacy, work-related fatigue, emotional distress, work characteristics, general health status, and basic demographic variables. The study should provide an assessment of whether principles of symptom self-management can be successfully applied to workplace problems and delivered in a group workshop format to reduce the disabling effects of chronic medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Workers with at least one chronic physical condition (> 6 months).
* Working full time (at least 20 hours per week).
* Able to read and speak in English language.

Exclusion Criteria:

* Impending retirement or major career change (next 12 months).
* Not available to attend group workshops after working hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2013-11; Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Work limitations | One year
  The Work Limitations Questionnaire (WLQ)(Lerner et al., 2003) is a 25-item self-report questionnaire that assesses the degree to which working individuals are experiencing limitations on-the-job due to their health problems and health-related productivity loss. The WLQ asks respondents to rate their level of difficulty or ability to perform specific job demands. Items are grouped into 4 scales: (1) time management; (2) physical demands; (3) mental-interpersonal demands; and (4) output demands.
Work engagement | One year
  The Utrecht Work Engagement Scale (UWES) (Demourati et al., 2001) is a 17-item self-report questionnaire that was designed to measure the degree to which employees have a sense of energetic and effective connection with their work activities (energy involvement) and see themselves as able to deal with the demands of their job (professional efficacy). Respondents rate their level of agreement with stated feelings about work on a 7-point likert scale from "never" to "always". Work engagement has been defined as a positive, fulfilling, work-related state of mind that is characterized by vigor, dedication, and absorption.

SECONDARY OUTCOMES:
Work fatigue | One year
  The Occupational Fatigue Exhaustion Recovery Scale (OFER) (Winwood et al., 2005) is a 20-item self-report questionnaire that assesses the degree to which job activities produce acute fatigue, deplete available energy, and reduce the ability to engage in pleasurable activities outside of work. Respondents rate their level of agreement on a 7-point likert scale from "completely disagree" to "completely agree".
Turnover intention | One year
  A 4-item scale developed by Kelloway and colleagues (1999) will be used to assess turnover intentions. The four questions are: "I am thinking about leaving this organization", "I am planning to look for a new job", "I intend to ask people about new job opportunities", and "I don't plan to be in this organization much longer". Each item is rated on a 5-point likert scale from "strongly disagree" to "strongly agree".
Job satisfaction | One year
  A 2-item scale developed from prior work by the researchers will be used to assess job satisfaction. The two questions are: "I like working for this company and expect to be here for another year or more" and "I would recommend this company to others".
Self-efficacy | One year
  A unique self-efficacy measure was developed for the project to be closely aligned with the content of the workshop program. Ten items were adapted from the Pain Self-efficacy Questionnaire (Nicholas, 2007) and ten items were taken from the Return-to-work Self Efficacy (RTWSE-19) scale (Shaw et al., 2011). The goal of the new measure is to assess worker confidence with respect to symptom management, job modification, communication, emotional coping, and obtaining needed support and assistance.
General health status | One year
  The Standard Form-36 (SF-36) (Ware et al., 1992) will be used to assess general health status. This is the most well-validated and frequently used measure of generic health status in health research. The SF-36 provides a single metric of health function regardless of diagnostic categories or illness classifications.
Sickness absence | One year
  Participants will be asked to recall the number of days in the past 6 months that they were absent from work because of their health. Self-report has been shown to be a viable and reasonably accurate method for assessing sickness absence days in studies of employee health (Short et al., 2009).
Healthcare utilization | One year
  Participants will be asked to recall the number and type of health care visits over the past 6 months using a standardized set of reporting options and prompts. Self-report has been shown to be a viable and reasonably accurate method for assessing health care utilization rates in studies of employee health (Short et al., 2009) and among individuals with chronic medical conditions (Lubeck & Hubert, 2005).

CONTACTS AND LOCATIONS:
Overall Officials: William S Shaw, Ph.D., Principal Investigator — Liberty Mutual Research Institute for Safety
Locations (4):
- United States (4):
  - Employer #3 (confidential), Worcester, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Hanover, New Hampshire
  - Employer #4 (Confidential), Hanover, New Hampshire
  - Employer #2 (confidential), Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be available to qualified researchers after data collection is complete

REFERENCES:
- [Background] Tveito TH, Shaw WS, Huang YH, Nicholas M, Wagner G. Managing pain in the workplace: a focus group study of challenges, strategies and what matters most to workers with low back pain. Disabil Rehabil. 2010;32(24):2035-45. doi: 10.3109/09638281003797398. Epub 2010 Sep 23. PMID 20860528
- [Background] Shaw WS, Tveito TH, Geehern-Lavoie M, Huang YH, Nicholas MK, Reme SE, Wagner G, Pransky G. Adapting principles of chronic pain self-management to the workplace. Disabil Rehabil. 2012;34(8):694-703. doi: 10.3109/09638288.2011.615372. Epub 2011 Oct 17. PMID 22004668
- [Background] Shaw WS, Tveito TH, Boot CR. Introduction to the special section: sustainability of work with chronic health conditions. J Occup Rehabil. 2013 Jun;23(2):157-61. doi: 10.1007/s10926-013-9448-7. PMID 23625029
- [Derived] Shaw WS, McLellan RK, Besen E, Namazi S, Nicholas MK, Dugan AG, Tveito TH. A Worksite Self-management Program for Workers with Chronic Health Conditions Improves Worker Engagement and Retention, but not Workplace Function. J Occup Rehabil. 2022 Mar;32(1):77-86. doi: 10.1007/s10926-021-09983-6. Epub 2021 May 13. PMID 33983524
- [Derived] Shaw WS, Besen E, Pransky G, Boot CR, Nicholas MK, McLellan RK, Tveito TH. Manage at work: a randomized, controlled trial of a self-management group intervention to overcome workplace challenges associated with chronic physical health conditions. BMC Public Health. 2014 May 28;14:515. doi: 10.1186/1471-2458-14-515. PMID 24885844